CLINICAL TRIAL: NCT03229174
Title: Evaluation of Brain Perfusion and Oxygenation in PD Patients With Neurogenic Orthostatic Hypotension: 4 Week Comparison of Droxidopa Versus Placebo
Brief Title: Brain Perfusion & Oxygenation in Parkinson's Disease With NOH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: William Ondo, MD (Other)
Collaborators: Lundbeck LLC (Industry)
Responsible Party: Sponsor-Investigator, William Ondo, MD, Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00013931
Record Dates: First submitted 2017-04-21; First posted 2017-07-25 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease; Neurogenic Orthostatic Hypotension
MeSH Terms: conditions — Parkinson Disease | interventions — Droxidopa; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention phase (Experimental): Droxidopa unforced titration dose (starting at 100mg by mouth TID) or matching placebo and titrated over 2 weeks up to maximum of 600 TID. Efficacy evaluation of given dose at week 4
  Interventions: Drug: Droxidopa; Drug: Placebo
- Open label extension phase (Other): All subjects allowed into a 4 week open label extension. Similar titration will start at 100mg Droxidopa three times a day (TID), but can be titrated up daily using the same dose escalation scale.
  Interventions: Drug: Droxidopa

INTERVENTIONS:
Drug: Droxidopa — Droxidopa initial dose 100mg TID, titrated in increments of 100mg every 24-48 hours to symptomatic response.
  Other Names: Northera
Drug: Placebo — Placebo (sugar pill)
  Other Names: Sugar pill
  Arms: Intervention phase

SUMMARY:
This is a double blind placebo controlled trial in Parkinson's disease (PD) patients with neurogenic orthostatic hypotension (NOH). Investigators hypothesize that the study drug (droxidopa) may improve cerebral perfusion more robustly than systemic BP, possibly by direct action within the CNS vasculature. This study is designed to determine if droxidopa improves cerebral perfusion measures in PD patients with NOH, in addition to peripheral BP measures and subjective responses.

DETAILED DESCRIPTION:
1. This is a double blind placebo controlled trial in PD patients with NOH. The controlled portion consists of two visits (baseline and week 4) and a phone call (week 2). An open label extension will include a phone call (week 6) and a final visit (week 8). Subjects will undergo a baseline assessment including continuous tilt table (10 minutes supine / 30 minutes at 70o / 10 minute supine) measurements of arteriole BP. Assessment will be done in the "on" state 1-3 hours after last dose and 1-3 hours after last meal. During both supine and standing positions, subjects will undergo a quantified transcranial cerebral ultrasound of the middle cerebral artery. A secondary analysis of the posterior circulation (basilar artery) will also be done when technically possible. An experienced technician will use a Spencer ST-3 Transcranial Doppler and MHz frequency probes (Spencer Technologies, Redmond WA), with ability to display all data in real time with M-mode and spectral waveform, depth of sample volume, size of sample volume, peak systolic and end diastolic velocities, pulsatility index and frequency of transducer. Cerebral oxygenation will be assessed throughout the tilt table with an FORE-SIGHT ELITE Oximetry System (CASMED) with FORE-SIGHT ELITE large advanced sensor. Mean/Max/Min vales will be analyzed. The tilt table BP and HR monitor with autonomic function will be recorded with a Task Force monitor from CNsystem. Subjective assessments will be done prior to the tilt table and will include demographics, general medical history, UPDRS, and the orthostatic hypotension questionnaire, and some gait analysis. We will also query their subjective "light headedness" throughout the tilt table test to determine for objective correlates.
2. Subjects will be titrated with droxidopa or matching placebo over two weeks using current guidelines. The dose will be held constant for the final two weeks and taken on the day of the week 4 visit. After a safety and dose determination call at two weeks, subjects will return at 4 weeks for an identical evaluation, along with clinical global impressions of change.
3. All subjects will be allowed into a 4 week open label extension. They will start titration at 100 mg droxidopa TID but can titrate up daily if preferred. After a safety call (week 6) they will return for a final tilt table/ultrasound perfusion study/oximetry study and subjective questionnaires. The patients will be provided two additional weeks medication to ensure a safe transition to purchased droxidopa if desired.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease patients with orthostatic hypotension (Systolic Blood Pressure drop of > 20 mm hg or Diastolic Blood Pressure drop of >10 mm hg measured at some point) within a month of inclusion.

Exclusion Criteria:

* Age >85
* Concurrent use of Midodrine
* Medical conditions that in the opinion of the investigator, might not allow for same completion of the study i.e. unstable angina, neoplasm, etc

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Cerebral perfusion | 8 weeks
  Cerebral perfusion measured by trans-cranial ultrasound of middle cerebral artery "supine and standing" delta.
Brain oxygenation | 8 weeks
  Brain oxygenation as measured by cerebral pulse oximetry device, delta between supine and standing

SECONDARY OUTCOMES:
Arteriole Blood Pressure | 8 weeks
  Change in arteriole BP (supine/standing) via tilt table
R-R variability | 8 weeks
  changes in autonomic influence on heart rate placebo vs drug
Orthostatic hypotension | 8 weeks
  Orthostatic hypotension scale
Assessment of Parkinson's disease symptoms | 8 weeks
  Movement disorder society- Unified parkinson disease rating scale (MDS-UPDRS)
Assessment of gait and falls | 8 weeks
  Timed Up and Go test

OTHER OUTCOMES:
Assessment of depressive symptoms | 8 weeks
  Beck Depression Inventory
Assessment of sleepiness | 8 weeks
  Epworth sleepiness scale (ESS)
Assessment of cognitive changes | 8 weeks
  Montreal cognitive assessment (MOCA)
Assessment of fatigue | 8 weeks
  Fatigue severity scale (FSS)
Participant impression of light-headedness | 8 weeks
  Subjective assessment of "light-headedness"

CONTACTS AND LOCATIONS:
Overall Officials: William Ondo, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No